CLINICAL TRIAL: NCT04080557
Title: Abdominal Aortic Aneurysm Patients Remain at Risk for Delirium on the Surgical Ward After Intensive Care Unit Dismissal
Status: Completed | Type: Observational
Sponsor: Amphia Hospital (Other)
Responsible Party: Principal Investigator, Joost Roijers, Principal Investigator, Amphia Hospital
Other Study IDs: 305213JR
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Delirium; AAA; Intensive Care Unit Delirium; Surgery--Complications; Surgery; Aortic Aneurysm, Abdominal
Keywords: delirium; intensive care unit; surgical ward; abdominal aortic aneurysm surgery
MeSH Terms: conditions — Delirium; Aortic Aneurysm, Abdominal | interventions — Surgical Procedures, Operative; Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AAA patients that went to the ICU postoperatively: An retrospective cohort study was conducted that included all patients treated electively for an abdominal aortic aneurysm (AAA) by open repair and patients undergoing emergency treatment for a ruptured AAA between 2013 and 2018.
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery — All patients treated electively for an abdominal aortic aneurysm (AAA) by open repair and patients undergoing emergency treatment for a ruptured AAA between 2013 and 2018.
  Other Names: Open abdominal aortic repair; Endovascular aortic repair

SUMMARY:
The incidence of delirium following open abdominal aortic aneurysm (AAA) surgery is significant, with incidence rates ranging from 12 to 33%. The occurrence of delirium on the surgical ward after intensive care unit (ICU) dismissal in AAA patients remains unclear. Differences in outcomes between a delirium on the ICU and a delirium on the surgical ward have not been previously investigated.

Delirium is a frequent complication in patients who underwent open AAA surgery. This study demonstrated that patients on the surgical ward remain at risk for developing a delirium after ICU dismissal. Physicians should therefore maintain a high level of awareness for delirium in AAA patients who return to the surgical ward after ICU dismissal. This simultaneously emphasises the necessity of delirium preventive measures and early recognition on the surgical ward in order to improve clinical outcomes.

DETAILED DESCRIPTION:
The incidence of delirium following open abdominal aortic aneurysm (AAA) surgery is significant, with incidence rates ranging from 12 to 33%. The occurrence of delirium on the surgical ward after intensive care unit (ICU) dismissal in AAA patients remains unclear. Differences in outcomes between a delirium on the ICU and a delirium on the surgical ward have not been previously investigated.

An observational cohort study was conducted that included all patients treated electively for an abdominal aortic aneurysm (AAA) by open repair and patients undergoing emergency treatment for a ruptured AAA between 2013 and 2018. The diagnosis of delirium was verified by a psychiatrist or geriatrician using the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria. Cox proportional hazards regression analysis was used to analyse 6- and 12-months survival rate.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated electively for an abdominal aortic aneurysm (AAA) by open repair and patients undergoing emergency treatment for a ruptured AAA between 2013 and 2018.

Exclusion Criteria:

* Patients that did not survive surgery
* Patients that did not go to the intensive care unit postoperatively.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 135 patients were included in the study. Of these, 72 were treated for a ruptured abdominal aortic aneurysm and 63 were treated electively with open aortic repair.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
the incidence of delirium | between january 2013 and december 2018
  The incidence of delirium on the ICU and on the ward

SECONDARY OUTCOMES:
mortality | 6 months and 12 months
  mortality divided by ICU delirium and ward delirium

OTHER OUTCOMES:
Length of hospital stay | Data on re-interventions, readmissions and survival were collected until February 2019.
  Length of hospital stay in days
Length of ICU stay | Data on re-interventions, readmissions and survival were collected until February 2019.
  Length of ICU stay in days
Reoperations | Data on re-interventions, readmissions and survival were collected until February 2019.
  Reoperations within 30 days after surgery
Complications | Data on re-interventions, readmissions and survival were collected until February 2019.
  Complications within 30 days after surgery
Discharge to a nursing home | Data on re-interventions, readmissions and survival were collected until February 2019.
  Discharge to a nursing home

CONTACTS AND LOCATIONS:
Overall Officials: Lijckle van der Laan, MD, PhD, Study Chair — Amphia hospital Breda, the Netherlands
Locations (1):
- Amphia hospital, Breda, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided